CLINICAL TRIAL: NCT01345006
Title: A Phase I/II, Open-Label, Multi-Center, Prospective Study to Determine the Safety and Tolerability of Sub-retinal Transplantation of Human Embryonic Stem Cell Derived Retinal Pigmented Epithelial (MA09-hRPE) Cells in Patients With Stargardt's Macular Dystrophy (SMD)
Brief Title: Sub-retinal Transplantation of hESC Derived RPE(MA09-hRPE)Cells in Patients With Stargardt's Macular Dystrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Institute for Regenerative Medicine (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7316-CL-0001; ACT SMD 01 MA09-hRPE (Other: Sponsor); ACT MA09-hRPE SMD-001 (Other: Sponsor)
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Stargardt's Macular Dystrophy
Keywords: juvenile macular dystrophy; SMD; fundus flavimaculatus
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MA09-hRPE (Experimental): Patients will undergo subretinal injection of MA09-hRPE
  Interventions: Biological: MA09-hRPE

INTERVENTIONS:
Biological: MA09-hRPE — Cohort 1 50,000 cells
  Cohort 2 100,000 cells
  Cohort 2a Better Vision 100,000 cells
  Cohort 3 150,000 cells
  Cohort 4 200,000 cells

SUMMARY:
This is a safety and tolerability trial to evaluate the effect of subretinal injection of human embryonic stem cell derived retinal pigment epithelium cells in patients with Stargardt's Macular Dystrophy (SMD).

DETAILED DESCRIPTION:
This study is a Phase I/II, open-label, non randomized, sequential, multi-center clinical trial. There will be 5 cohorts, the 4 low vision cohorts will contain 3 patients, the better vision cohort will contain 4 patients. The enrolled cohorts will be as follows:

Three SMD patients- 50,000 MA09-hRPE cells transplanted

Three SMD patients- 100,000 MA09-hRPE cells transplanted

Four Better Vison SMD patients- 100,000 MA09-hRPE cells transplanted

Three SMD patients- 150,000 MA09-hRPE cells transplanted

Three SMD patients- 200,000 MA09-hRPE cells transplanted

Patients will be enrolled sequentially, and within each cohort of 3 patients, each patient's clinical course over the first 6 weeks following cell transplantation will be reviewed by an independent (DSMB) before enrollment is opened for the next 2 patients. A full safety assessment of all 3 patients in each cohort will be made by the DSMB when the 3rd patient in each cohort completes 4 weeks of follow-up, and before the first patient in the next cohort receives a cell transplant. The exception is the better vision group where all patients may be enrolled once DSMB approval has been received.

Each cohort will be enrolled sequentially in turn, with the exception of the better vision cohort which may be enrolled in parallel with the other cohorts.

The day of the cell implantation will be Day 0, and patients will remain in the study until the last visit at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female over 18 years of age.
* Clinical diagnosis of advanced SMD.
* If known, the patient's genotype will be recorded in the medical history, if unknown, patient will allow for the submission of a sample for genotyping.Clinical findings consistent with SMD.
* The visual acuity of the eye to receive the transplant will be no better than 20/400. The visual acuity of the eye in the better vision cohort to receive the transplant will be no better than 20/100.
* The visual acuity of the eye that is not to receive the transplant will be no better than 20/400 for the worse vision patients and no worse than 20/100 for the better vision patients.
* Peripheral visual field constriction documented on standard kinetic visual field testing.
* Electrophysiological findings consistent with SMD.
* Medically suitable to undergo vitrectomy and subretinal injection.
* Medically suitable for general anesthesia or waking sedation, if needed.
* Medically suitable for transplantation of an embryonic stem cell line:
* Normal serum chemistry (sequential multi-channel analyzer 20 [SMA- 20]) and hematology (complete blood count [CBC], prothrombin time [PT], and activated partial thromboplastin time [aPTT]) screening tests.
* Negative urine screen for drugs of abuse.
* Negative human immunodeficiency virus (HIV), hepatitis B (HBV), hepatitis C (HCV) serologies.
* No history of malignancy,with the exception of successfully treated basal cell or squamous cell carcinoma of the skin.
* Negative cancer screening within previous 6 months:
* complete history & physical examination;
* dermatological screening exam for malignant lesions;
* negative fecal occult blood test & if over age 50 years, negative colonoscopy within previous 7 years;
* negative chest roentgenogram (CXR);
* normal CBC & manual differential;
* negative urinalysis (U/A);
* normal thyroid exam;
* if male, normal testicular examination; if over age 40, digital rectal examination (DRE) and prostate specific antigen (PSA);
* if female, normal pelvic examination with Papanicolaou smear; and
* if female, normal clinical breast exam and if 40 years of age or older, negative mammogram.
* If female and of childbearing potential, willing to use two effective forms of birth control during the study.
* If male, willing to use barrier and spermicide contraception during the study.
* Willing to defer all future blood, blood component or tissue donation. -Able to understand and willing to sign the informed consent.

Exclusion Criteria:

* History of malignancy,with the exception of successfully treated basal cell or squamous cell carcinoma of the skin.
* History of myocardial infarction in previous 12 months.
* History of diabetes mellitus.
* Any immunodeficiency.
* Any current immunosuppressive therapy other than intermittent or low dose corticosteroids.
* Serologic evidence of infection with Hepatitis B, Hepatitis C, or HIV.
* Current participation in any other clinical trial.
* Participation within previous 6 months in any clinical trial of a drug by ocular or systemic administration.
* Any other sight-threatening ocular disease.
* Any chronic ocular medications.
* Any history of retinal vascular disease (compromised blood-retinal barrier.
* Glaucoma.
* Uveitis or other intraocular inflammatory disease.
* Significant lens opacities or other media opacity.
* Ocular lens removal within previous 3 months.
* If female, pregnancy or lactation.
* Any other medical condition, which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromises patient safety, or interferes with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-06-16 (Actual); Primary Completion 2015-08-10 (Actual); Study Completion 2015-08-10 (Actual)

PRIMARY OUTCOMES:
The safety and tolerance of transplantation of hESC-derived RPE cells MA09-hRPE | 12 months
  The transplantation of hESC-derived RPE cells MA09-hRPE will be considered safe and tolerated in the absence of:
  * Any grade 2 (NCI grading system) or greater adverse event related to the cell product
  * Any evidence that the cells are contaminated with an infectious agent
  * Any evidence that the cells show tumorigenic potential
Safety Assessments | 12 months
  * Adverse Event and Serious Adverse Event assessment
  * Clinical monitoring
  * Serial vital signs
  * Clinical laboratory tests
  * Directed ophthalmological monitoring
  * Monitoring of RPE cells acceptance/integrity/rejection
  * Monitoring of local and systemic infection
  * Monitoring of tumorigenic cell transformation

SECONDARY OUTCOMES:
Evidence of successful engraftment | 12 months
  Evidence of successful engraftment will consist of:
  * Structural evidence (OCT imaging, fluorescein angiography, autofluorescence photography, slit-lamp examination with fundus photography) that cells have been implanted in the correct location
  * Electroretinographic evidence (mfERG) showing enhanced activity in the implant location

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Institute for Regenerative Medicine
Locations (3):
- United States (3):
  - Jules Stein Eye Institute, UCLA School of Medicine, Los Angeles, California
  - Bascom Palmer Eye institute, Miami, Florida
  - Wills Eye Institute-Mid Atlantic Retina, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Davis JL. The Blunt End: Surgical Challenges of Gene Therapy for Inherited Retinal Diseases. Am J Ophthalmol. 2018 Dec;196:xxv-xxix. doi: 10.1016/j.ajo.2018.08.038. Epub 2018 Sep 5. PMID 30194931
- [Derived] Schwartz SD, Regillo CD, Lam BL, Eliott D, Rosenfeld PJ, Gregori NZ, Hubschman JP, Davis JL, Heilwell G, Spirn M, Maguire J, Gay R, Bateman J, Ostrick RM, Morris D, Vincent M, Anglade E, Del Priore LV, Lanza R. Human embryonic stem cell-derived retinal pigment epithelium in patients with age-related macular degeneration and Stargardt's macular dystrophy: follow-up of two open-label phase 1/2 studies. Lancet. 2015 Feb 7;385(9967):509-16. doi: 10.1016/S0140-6736(14)61376-3. Epub 2014 Oct 15. PMID 25458728
- [Derived] Schwartz SD, Hubschman JP, Heilwell G, Franco-Cardenas V, Pan CK, Ostrick RM, Mickunas E, Gay R, Klimanskaya I, Lanza R. Embryonic stem cell trials for macular degeneration: a preliminary report. Lancet. 2012 Feb 25;379(9817):713-20. doi: 10.1016/S0140-6736(12)60028-2. Epub 2012 Jan 24. PMID 22281388
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/patientStudySearch.aspx?RID=;;;7316-CL-0001
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217491&parentIdentifier=7316-CL-0001&attachmentIdentifier=980e257a-46d6-47c2-8188-165bb8b8be73&fileName=7316-CL-0001_0004_Plain_language_summary.pdf&versionIdentifier=